CLINICAL TRIAL: NCT00092066
Title: A 15-Week, Double-Blind, Randomized, Active-Controlled, Multi-Center Study With 24-Week Extension to Evaluate the Safety, Tolerability, Efficacy of Alendronate 70 mg Plus Vitamin D3 2800 IU Combination Tablet in Men and Postmenopausal Women With Osteoporosis
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of an Investigational Drug and Dietary Supplement in Men and Postmenopausal Women With Osteoporosis (0217A-227)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0217A-227; 2004_020
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis; Vitamin D Deficiency
MeSH Terms: conditions — Osteoporosis; Vitamin D Deficiency | interventions — Alendronate; Cholecalciferol; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0217A, alendronate sodium (+) cholecalciferol / Duration of Treatment: 15 weeks

SUMMARY:
The purpose of this study is to test the safety, tolerability and effectiveness of an investigational drug and dietary supplement to reduce the risk of vitamin D insufficiency and deficiency during the treatment of osteoporosis in men and postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Men or postmenopausal women who are osteoporotic

Exclusion Criteria:

* Vitamin D deficiency
* Other disease of bone or mineral metabolism
* Digestive disease causing malabsorption
* Other significant medical conditions that are not adequately treated

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 717 (Actual)
Dates: Start 2003-09-24 (Actual); Primary Completion 2004-05-01 (Actual); Study Completion 2004-05-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Vitamin D insufficiency (defined as serum 25-hydroxyvitamin levels <15 ng/mL) after 15 weeks of treatment.

SECONDARY OUTCOMES:
Proportion of patients with vitamin D deficiency (serum 25-hydroxyvitamin D levels <9 ng/mL) after 15 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Recker R, Lips P, Felsenberg D, Lippuner K, Benhamou L, Hawkins F, Delmas PD, Rosen C, Emkey R, Salzmann G, He W, Santora AC. Alendronate with and without cholecalciferol for osteoporosis: results of a 15-week randomized controlled trial. Curr Med Res Opin. 2006 Sep;22(9):1745-55. doi: 10.1185/030079906x120913. PMID 16968578